CLINICAL TRIAL: NCT00311766
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Response Study of the Safety and Efficacy of Thymosin Beta 4 in the Treatment of Patients With Epidermolysis Bullosa
Brief Title: A Phase 2 Study on Effect of Thymosin Beta 4 on Wound Healing in Patients With Epidermolysis Bullosa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patient availability and expiration of study drug
Sponsor: RegeneRx Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSEB; 0003031 (Other: FDA Office of Orphan Product Development (OOPD))
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; cutaneous wound-healing; chronic wound-healing; Thymosin Beta 4; laminin-5
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo comparator gel does not contain any active drug. Topical administration of 0.0% Thymosin Beta 4 gel, once a day (qd) up to 56 days
  Interventions: Drug: Placebo
- 2 (Active Comparator): Topical Administration of 0.01%, 0.03%, and 0.1% Thymosin Beta 4 gel once a day (qd) up to 56 days
  Interventions: Drug: Thymosin Beta 4

INTERVENTIONS:
Drug: Thymosin Beta 4 — Topical administration, 0.01%, 0.03%, and 0.1% Thymosin Beta 4 gel, qd up to 56 days
  Arms: 2
Drug: Placebo — Topical administration, 0.00% Thymosin Beta 4 gel qd up to 56 days
  Arms: 1

SUMMARY:
The purpose of this study is to investigate a treatment to enhance the healing of acute and chronic nonhealing cutaneous wounds, such as the erosions experienced by patients with Epidermolysis Bullosa (EB), by the known activity of thymosin beta 4 (Tβ4). Funding Source - FDA Office of Orphan Product Development (OOPD).

DETAILED DESCRIPTION:
EB is a group of genetic diseases characterized by skin-blistering and lesion-formation after minor trauma to the skin. This family of disorders, most of which are inherited, range in severity from mild to the severely disabling and life-threatening. Tβ4 is a synthetically-produced copy of a naturally-occurring 43 amino acid peptide that has wound healing and anti-inflammatory properties and can up-regulate the expression of laminin-5.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent form signed by the patient or patient's legal representative; also, if the patient is under the age of majority but capable of providing assent, signed assent from the patient
* Diagnosis of junctional or dystrophic EB.
* Patients who present with Hallopeau-Siemens subtype may be enrolled.
* At least one active, unroofed EB erosion on the limb or on the trunk.
* Lesion size 5 to 50 cm2, inclusive.
* Stable lesion present for 14-60 days before enrollment.
* More that one member in a family can be enrolled as long as that member is treated to a different cohort with an assurance that the study medication will not be shared.
* No clinically significant abnormalities (Grade 2 or higher on the National Cancer Institute [NCI] toxicity scale) on Screening laboratory tests, except for the following specific laboratory threshold result: albumin must be 2 g/dL or higher; hemoglobin must be 8 g/dL or higher.

Exclusion Criteria:

* Clinical evidence of local infection of the index (targeted) lesion.
* Use of any investigational drug within the 30 days before enrollment.
* Use of immunotherapy or cytotoxic chemotherapy within the 60 days before enrollment.
* Use of systemic or topical steroidal therapy within the 30 days before enrollment.Inhaled steroids are allowed.
* Use of systemic antibiotics within the 7 days before enrollment.
* Current or former malignancy.
* Arterial or venous disorder resulting in ulcerated wounds.
* Diabetes mellitus.
* Pregnancy or breastfeeding during the study. (A serum pregnancy test will be performed at Screening for female patients of childbearing potential.)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2010-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Crockford, Study Director — RegeneRx Biopharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In:22 February 2006; Last Patient In: 6 July 2010 Locations: Medical Centers
Pre-assignment Details: No wash out or run-in periods in this study
Groups:
- Placebo: Topical administration of placebo gel, 0% Thymosin Beta 4, qd up to 56 days
  Placebo : Topical administration, 0.00% qd up to 56 days
- Thymosin Beta 4: Topical administration of 0.01%, 0.03%, and 0.1% Thymosin Beta 4 gel, qd up to 56 days
  Thymosin Beta 4 : Topical administration, 0.01%, 0.03%, and 0.1% gel, qd up to 56 days
Period: Overall Study
Arm/Group | Placebo | Thymosin Beta 4
Started | 8 | 22
Completed | 8 | 17
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Thymosin Beta 4 | Total
Number analyzed (Participants) | 8 | 22 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 12 | 16
  Between 18 and 65 years | 4 | 10 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 6 | 14 | 20
Region of Enrollment [Number; unit: participants]
  United States | 8 | 22 | 30

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Whose Wounds Have Healed
Description: Wound healing means that the wound has closed without any drainage
Time Frame: 56 days
Population: The population for efficacy analysis will be the Full Analysis (FA) population. The FA analysis included all patients who were randomized and received at least one dose of study medication and who had at least one baseline efficacy parameter recorded.
Measure: Number; unit: participants
Arm/Group | Placebo | Thymosin Beta 4
Number analyzed (Participants) | 8 | 22
participants | 5 | 8
Statistical Analysis 1: Comparison: Placebo vs Thymosin Beta 4; The primary population was the Full Analysis(FA)population. The FA population included all patients who were randomized and received at least one dose of study medication and who had at least one baseline efficacy parameter recorded; Test type: Superiority or Other; p > 0.05, Fisher Exact; ANCOVA = 0.80

2. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: 70 days
Population: The population for safety analysis included all patients who were randomized and received at least one dose of study medication and had at one safety parameter recorded.
Measure: Number; unit: Participants
Arm/Group | Placebo | Thymosin Beta 4
Number analyzed (Participants) | 8 | 22
Participants
  Adverse Events | 0 | 1
  Serious Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected within 70 days
Arm/Group | Placebo | Thymosin Beta 4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/22
Other Adverse Events (participants affected / at risk) | 0/8 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Thymosin Beta 4 (N=22)
cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Cellulitis was resolved in 27 days

LIMITATIONS AND CAVEATS:
Early termination of the study leading to randomizing 30 of the 36 participants planned. This was due to the small pool of participants and therefore resulting in low availability of eligible participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less